CLINICAL TRIAL: NCT02360124
Title: Randomized Clinical Trial on Preventing and Arresting Dental Root Surface Caries Using Silver Diamine Fluoride Solution in Community-dwelling Older Adults
Brief Title: Preventing and Arresting Dental Root Surface Caries in Community-dwelling Older Adults
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UW11-120
Record Dates: First submitted 2014-11-17; First posted 2015-02-10 (Estimated); Results first posted 2016-05-19 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-06

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — silver diamine fluoride; Water

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- control (Placebo Comparator): instructions on oral hygiene (OHI) tailored to the individual's condition will be given, and a tube of toothpaste containing 1,000 ppm fluoride (the most popular type of adult toothpaste in the Hong Kong market) will be provided. The OHI and provision of toothpaste will be repeated at 6-month intervals. In addition, distilled water as placebo with a bitter flavor added (to mimic the bitter metallic taste of SDF) will be painted onto all exposed tooth root surfaces using a small disposable brush. This procedure will be repeated after 12 and 24 months.
  Interventions: Other: Water as placebo
- silver diammine fluoride (Experimental): the subjects will receive the same intervention as those provided to subjects in the control group except that a 38% SDF solution (Saforide, Toyo Seiyaku Kasei Co. Ltd, Osaka, Japan) instead of the placebo solution will be painted onto the exposed tooth root surfaces. This treatment will be repeated after 12 and 24 months.
  Interventions: Drug: silver diammine fluoride
- silver diammine fluoride and KI (Active Comparator): the subjects will receive the same treatment as those provided to subjects in the control group except that a 38% SDF solution instead of the placebo solution will be painted onto the exposed tooth root surfaces and followed by painting of a saturated potassium iodide solution. This treatment will be repeated after 12 and 24 months.
  Interventions: Drug: silver diammine fluoride; Other: saturated potassium iodide solution

INTERVENTIONS:
Drug: silver diammine fluoride — topical application of the SDF solution onto tooth root surfaces
  Other Names: SDF
  Arms: silver diammine fluoride; silver diammine fluoride and KI
Other: Water as placebo — topical application of water as a placebo in the control arm
  Other Names: Water
  Arms: control
Other: saturated potassium iodide solution — topical application of SDF solution followed by KI solution onto tooth root surfaces
  Other Names: KI
  Arms: silver diammine fluoride and KI

SUMMARY:
This study is a randomized clinical trial lasting for 30 months. A total of 300 subjects will be recruited from social centres for elders located in different districts in Hong Kong. Baseline clinical examination will be conducted by a single calibrated examiner in the social centres using an intra-oral LED light, mouth mirrors and probes. Subjects will be randomly allocated into the three study groups and receive interventions accordingly. Follow-up examinations at 6-month intervals will be carried out to assess the clinical outcomes, i.e. whether new root caries has developed and whether the active root caries found at baseline have become arrested (remineralized and hardened) or not. Photographs of the arrested lesions will be taken to assess their colour. Results of this study will provide the much needed evidence to guide the dental professionals in Hong Kong and worldwide in deciding on the most appropriate intervention for the prevention and treatment of this common dental disease of the older adults.

DETAILED DESCRIPTION:
The primary and secondary outcome of this study was new root caries and arrested root caries. A root surface with new caries experience was recorded when a root surface which was sound at baseline was found to have a carious lesion or a filling at a follow-up examination. Arrested root caries was recorded when the active root caries found at baseline changed into inactive root caries at follow-up. The status of each root surface was recorded using the codes recommended by the International Caries Detection and Assessment System (ICDAS Ⅱ) Coordinating Committee in 2009. Color of the arrested root caries lesion was classified into one of four types according to PANTONE® color plates placed next to the lesion (Fig 1), namely yellow (7401U), light brown (1245U), dark brown (4635U), and black (Black U).

A mean root caries increment of around 0.8 root surface per year of control group was reported in a previous clinical trial conducted in Hong Kong. Thus, in this study, a 30-month increment of 2 new decayed root surfaces was anticipated. The ratio of the mean to the standard deviation of the root caries increment was expected to be around 1:1.5. In order to show that a 50% difference in mean caries increment between the highest and the lowest values in the three groups was statistically significant at a 5% significance level and at an 80% power, 80 subjects in each group was required. Allowing for a drop-out rate of 25% over 30 months, a total of 300 subjects (100 in each group) were needed.

ELIGIBILITY:
Inclusion criteria:

* have at least 5 teeth with exposed root surfaces and not indicated for extraction, and
* living in the community and have self-care ability for normal daily activities.

Exclusion Criteria:

* have life-threatening or serious health problems,
* have cognitive problems in communication or in receiving oral hygiene instructions
* have salivary gland diseases or received radiotherapy in the head and neck region.

Ages: 56 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2012-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward CM Lo, BDS, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No
We consider individual request case by case

REFERENCES:
- [Derived] Li R, Lo ECM, Liu BY, Wong MCM, Chu CH. Randomized Clinical Trial on Preventing Root Caries among Community-Dwelling Elders. JDR Clin Trans Res. 2017 Jan;2(1):66-72. doi: 10.1177/2380084416668491. Epub 2016 Sep 28. PMID 30938645

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: instructions on oral hygiene (OHI) tailored to the individual's condition will be given, and a tube of toothpaste containing 1,000 ppm fluoride (the most popular type of adult toothpaste in the Hong Kong market) will be provided. The OHI and provision of toothpaste will be repeated at 6-month intervals. In addition, distilled water with a bitter flavor added (to mimic the bitter metallic taste of SDF) will be painted onto all exposed tooth root surfaces using a small disposable brush. This procedure will be repeated after 12 and 24 months.
  Water as placebo: topical application of water as a placebo in the control arm
Period: Overall Study
Arm/Group | Control | Silver Diammine Fluoride | Silver Diammine Fluoride and KI
Started | 108 | 107 | 108
Completed | 80 | 95 | 82
Not Completed | 28 | 12 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Silver Diammine Fluoride | Silver Diammine Fluoride and KI | Total
Number analyzed (Participants) | 108 | 107 | 108 | 323
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 12 | 9 | 44
  >=65 years | 85 | 95 | 99 | 279
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.1 (6.7) | 72.4 (6.2) | 72.7 (5.8) | 72.1 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 83 | 84 | 253
  Male | 22 | 24 | 24 | 70
Race/Ethnicity, Customized [Number; unit: participants]
  Chinese | 108 | 107 | 108 | 323
Region of Enrollment [Number; unit: participants]
  China | 108 | 107 | 108 | 323

OUTCOME MEASURES:

1. Primary Outcome: Number of New Tooth Root Caries Lesions
Description: the number of new tooth root caries lesions, i.e. tooth roots that have changed from sound at baseline to decayed at the evaluation examination will be counted in the clinical examination
Time Frame: 30 months
Measure: Mean (Standard Error); unit: new carious root surfaces
Arm/Group | Control | Silver Diammine Fluoride | Silver Diammine Fluoride and KI
Number analyzed (Participants) | 80 | 95 | 82
new carious root surfaces | 1.1 (0.16) | 0.43 (0.09) | 0.56 (0.11)

2. Secondary Outcome: Proportion of Inactive Root Caries Lesions
Description: the proportion of active tooth root caries lesions at baseline that has changed to inactive root caries lesions at the evaluation examination will be calculated. The calculation is to divide the number of caries lesions that have changed status from active to inactive (assessed in clinical examination) by the number of active caries lesions found at baseline
Time Frame: 30 months
Population: The participants were the active root caries lesions found at baseline in each group.
Measure: Number; unit: percentage of inactive root caries
Arm/Group | Control | Silver Diammine Fluoride | Silver Diammine Fluoride and KI
Number analyzed (Participants) | 20 | 40 | 40
percentage of inactive root caries | 45.0 | 90.0 | 92.5

ADVERSE EVENTS:
Time Frame: 30 months
Arm/Group | Control | Silver Diammine Fluoride | Silver Diammine Fluoride and KI
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/107 | 0/108
Other Adverse Events (participants affected / at risk) | 0/108 | 0/107 | 0/108

LIMITATIONS AND CAVEATS:
It should be noted that the water in Hong Kong is fluoridated at an optimal concentration of 0.5 ppm, and whether SDF or SDF/KI is effective among elders living in non-fluoridated areas needs to be investigated in future clinical studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No